CLINICAL TRIAL: NCT02837029
Title: Phase I/Ib Study of Nivolumab in Combination With Therasphere (Yttrium-90) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Nivolumab and Yttrium Y 90 Glass Microspheres in Treating Patients With Advanced Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 16I01; STU00203003 (CTRP (Clinical Trial Reporting Program)); NU 16I01 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-01001 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-07-15; First posted 2016-07-19 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Stage IIIA Hepatocellular Carcinoma; Stage IIIB Hepatocellular Carcinoma; Stage IIIC Hepatocellular Carcinoma; Stage IVA Hepatocellular Carcinoma; Stage IVB Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (yttrium Y 90 glass microspheres, nivolumab) (Experimental): Patients receive yttrium Y 90 glass microspheres IA. Approximately 4 weeks after yttrium Y 90 glass microspheres treatment, patients receive nivolumab IV over 30-60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Radiation: Yttrium Y 90 Glass Microspheres

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Yttrium Y 90 Glass Microspheres — Given IA
  Other Names: TheraSphere

SUMMARY:
The purpose of this study is to identify maximum tolerated dose (MTD), that is, the highest dose of the study drug nivolumab that does not cause unacceptable side effects, for combination treatment of nivolumab and yttrium Y 90 glass microspheres (Y-90). Also, to evaluate the efficacy (the effect of drug on your tumor) and the tolerability (the effect of the drug on your body) of nivolumab, when given with standard of care Y-90 (Therasphere). Nivolumab is currently Food and Drug Administration (FDA) approved for other cancers, but has not yet been investigated in advanced or refractory hepatocellular carcinoma. Nivolumab is an antibody (a human protein that sticks to a part of the tumor and/or immune cells) designed to allow the body's immune system to work against tumor cells. Y-90 is currently FDA approved for the treatment of hepatocellular carcinomas, but has not yet been investigated in combination with nivolumab for this disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify MTD of nivolumab for combination treatment of nivolumab and Y-90 in this population.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients with objective response rate (ORR) (according to Response Evaluation Criteria in Solid Tumors [RECIST] criteria) to the combination treatment of nivolumab with Y-90.

II. To evaluate the proportion of patients alive and progression free at 24 weeks in the described population.

III. To evaluate the toxicities (according to the National Comprehensive Cancer Network [NCCN] Common Terminology Criteria for Adverse Events [CTCAE] version (v)4.03) and tolerability of nivolumab and Y-90 in patients with advanced hepatocellular carcinoma IV. To determine the disease control rate (DCR) to the combination of nivolumab and Y-90 at 24 months from the start of nivolumab treatment.

TERTIARY OBJECTIVES:

I. Programmed cell death 1 ligand 1 (PD-L1) protein on tumor cells and the expression levels of other markers of inflammatory/immune signature that may include but not be limited to programmed cell death protein 1 (PD-1), tumor necrosis factor receptor superfamily, member 4 (OX40), cluster of differentiation (CD) 73, CD39, T cell immunoglobulin and T-cell immunoglobulin and mucin-domain containing-3 (TIM3), glucocorticoid-induced tumour necrosis factor receptor (GITRL), cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), CD3, CD4, CD8, CD45RO, forkhead box P3 (FOXP3), and granzyme by immunohistochemistry (IHC) and/or flow cytometry will be evaluated.

II. Whole exome sequencing and computational analyses will be performed to assess mutanome and immunome (subpopulations of immune cells).

III. Change in clonal burden landscape of various mutanome and immunome will be analyzed to investigate its correlation with treatment response or development of resistance to treatment.

OUTLINE: This is a phase I, dose-escalation study of nivolumab followed by a phase Ib study.

Patients receive yttrium Y 90 glass microspheres intraarterially (IA). Approximately 7-14 days after Y-90 administration. A delay of 4 weeks will be permitted in case of toxicity. After yttrium Y 90 glass microspheres treatment, nivolumab will be administered intravenously (IV) over approximately 60 minutes every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent.

After completion of study treatment, patients are followed up 30 days after the last dose of nivolumab and again at 100 days after discontinuing study drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of hepatocellular carcinoma (HCC) confirmed by American Association for Study of Liver Diseases (AASLD) guidelines with a Childs-Pugh score of A or B (but, =< Childs score B8)

  * NOTE: If the patient does not have histological confirmation of disease by biopsy, diagnosis of HCC must be documented with approval by a tumor board or other multidisciplinary conference
* Patients must have at least 1 lesion that is measurable using RECIST guidelines.

NOTE: A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable per RECIST, and has clearly progressed.

NOTE: For patients with infiltrative disease, evaluable disease needs to be confirmed by pathology if RECIST measurements cannot be made.

* Patients must have advanced disease that is not amenable to transplant or resection
* Patients may be treatment naive or have received any number of prior therapies

  * NOTE: Prior immunotherapy is contraindicated and not permitted
* Patients with chronic hepatitis B are eligible as long as they have evidence of ongoing viral replication (detectable hepatitis B surface antigen [HBsAg], hepatitis B envelope antigen [HBeAg], or hepatitis B virus [HBV] deoxyribonucleic acid [DNA]); they must have HBV DNA viral load < 100 IU/mL at screening; in addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy; if not on antiviral therapy at screening, then the subject must initiate treatment per regional standard of care guidelines at the time of consent; both HBeAg positive and negative patients will be included
* Patients positive for hepatitis C are permitted if controlled with medication, in the opinion of the investigator
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patients must have adequate organ function within 14 days prior to registration as determined by:

  * Hematological (without growth factor support)
  * Hemoglobin >= 8.5 g/dL (without the use of growth factors)
  * Absolute neutrophil count (ANC) >= 1000
  * Platelet count >= 50 x 10^9/L (without use of growth factors [ie., interleukin 11 (oprelvekin)])
  * Prothrombin time (PT)/international normalized ratio (INR) =< 2.3 or PT =< 6 seconds above control
  * NOTE: Abnormal PT/INR may be considered, with documented principal investigator (PI) approval, if it is due to the use of anticoagulants; for such patients, a normal PT/INR must be available from before the start of anticoagulation treatment
* Renal

  * Calculated creatinine clearance (CrCl) or 24-hour urine CrCl > 50 mL/min (Cockcroft-Gault formula will be used to calculate CrCl)
* Hepatic

  * Serum bilirubin =< 3 times the upper limit of normal (ULN)
  * Aspartate aminotransaminase (AST) and alanine aminotransaminase (ALT) =< 5 times ULN
* Serum electrolytes

  * Lipase =< 1.5 times ULN
  * Amylase =< 1.5 times ULN
* Potassium, sodium, magnesium, and calcium (corrected for serum albumin) =< grade 1 or within the institutional ranges of normal; if clinically appropriate, electrolytes may be corrected and values reassessed prior to enrollment
* Females of childbearing potential (FOCBP), and non-sterilized males who are sexually active must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective; they must also refrain from egg and/or sperm cell donation and breastfeeding for 90 days after the final dose of investigational product(s)

  * FOCBP are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause)
  * Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab plus 5 half-lives of nivolumab (19 weeks) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post-treatment completion.
  * Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with nivolumab plus 5 half-lives of the study drug (19 weeks) plus 90 days (duration of sperm turnover) for a total of 31 weeks post-treatment completion
* FOCBP must have a negative pregnancy test within 7 days prior to registration

  * Note: FOCBP will have to have repeat pregnancy test within 24 hours of starting nivolumab, scheduled for cycle 1 day 1
* Subjects must provide archived tumor specimens for correlative biomarker studies if sufficient tissue is available; a fresh biopsy is not required
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients must not have had prior treatment with nivolumab or any other PDL1 or PD-1 antagonists
* Patients must not have a history of severe allergic reactions (i.e., grade 4 allergy, anaphylactic reaction from which the subject did not recover within 6 hours of institution of supportive care) to any unknown allergens or any components of the nivolumab formulations
* Patients diagnosed or treated for malignancy other than HCC are not eligible unless they meet one of the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for >= 3 years before registration and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded; these include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn's
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome
  * NOTE: Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients with renal failure currently requiring dialysis of any kind are not eligible
* Patients with untreated central nervous system (CNS) metastatic disease (including spinal cord and leptomeningeal disease) are excluded

  * Note: Subjects with previously treated CNS metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management are permitted to enroll
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study, is excluded
* Receipt of any investigational therapy is not permitted within 28 days prior to the first dose of nivolumab
* Any concurrent chemotherapy, biologic or hormonal therapy for cancer treatment is not permitted within 28 days of registration

  * Note: Prior immunotherapy is not permitted
  * Note: Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable
* Patients with exposure to prior immunotherapy are not eligible
* Patients are ineligible if they have unresolved toxicities from prior anticancer therapy, defined as having not resolved to National Cancer Institute (NCI) CTCAE version 4.03 grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria

  * Note: Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (eg, hearing loss) after consultation with the PI and Northwestern University (NU) Quality Assurance Monitor (QAM)
* Radiation therapy is not permitted within 14 days of registration
* Live vaccines are not permitted within 28 days of study registration
* No systemic glucocorticoids will be permitted within 48 hours prior to study registration

  * Note: Topical steroids, bronchodilators and local steroid injections are permitted if clinically required
* Patients with cardiac disease defined as one of the following are not eligible:

  * Congestive heart failure > class II New York Heart Association (NYHA)
  * Unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months)
  * Myocardial infarction within the past 6 months
* Patients with cardiac ventricular arrhythmias requiring anti-arrhythmic therapy are not eligible
* Patients with known human immunodeficiency virus (HIV) infection are not eligible
* Patients must not have elevated lung shunting precluding treatment with Y-90
* Patients who have had major surgery within 4 weeks prior to registration are not eligible
* Patients who have active clinically serious infection > CTCAE grade 2 are not eligible
* Patients with a history of gastrointestinal bleeding (GIB) within 6 weeks prior to registration are not eligible
* Patients with prior transplant of any kind are not eligible
* Known or suspected allergy to nivolumab or any agent given in the course of this trial is not permitted
* Patients may not be pregnant or lactating at study registration
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension (defined as > 150/90) that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
  * Active alcohol use, drug use, or a psychiatric disease that would, in the opinion of the PI or a sub-investigator (sub-I), prevent the subject from complying with the study protocol and/or endanger the subject during their participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07; Primary Completion 2019-07-17 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Kalyan, MBBS, FRACP, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on July 25th, 2016 with goal of 40 patients. The first patient started treatment Sep. 12, 2016. The study design for Phase 1 was 3 + 3 dose escalation. Accrual was suspended on June 7, 2019 for review of DLT data for dose Level 2 of Phase 1. The study closed Jun. 2, 2020 due to funding issues and Phase 1b never opened.
Groups:
- Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks): Nivolumab was administered at 80mg as an intravenous infusion over 30 minutes (-5 minutes / +15 minutes) every 2 weeks (Day 1 & 15 of each cycle, 1 Cycle = 28 days). Courses repeated every cycle in the absence of disease progression or unacceptable toxicity.
  Correlatives studies: Peripheral lymphocyte analysis, and analysis for PD-K1, PD-1, CD8+, and CD4+ tumor infiltrating lymphocytes.
- Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks): Nivolumab was administered at 240mg as an intravenous infusion over 30 minutes (-5 minutes / +15 minutes) every 2 weeks (Day 1 & 15 of each cycle, 1 Cycle = 28 days). Courses repeated every cycle in the absence of disease progression or unacceptable toxicity.
  Correlatives studies: Peripheral lymphocyte analysis, and analysis for PD-K1, PD-1, CD8+, and CD4+ tumor infiltrating lymphocytes.
- Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks): The maximum tolerated dose of nivolumab was planned to be administered in patients recruited to Phase 1b, as an intravenous infusion over 30 minutes (-5 minutes / +15 minutes) every 2 weeks (Day 1 & 15 of each cycle, 1 Cycle = 28 days). Courses would repeat every cycle in the absence of disease progression or unacceptable toxicity.
  Correlatives studies: Peripheral lymphocyte analysis, and analysis for PD-K1, PD-1, CD8+, and CD4+ tumor infiltrating lymphocytes.
  Phase 1b never opened to accrual due to funding issues.
Period: Screening
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Started | 15 | 12 | 0
Completed | 8 | 9 | 0
Not Completed | 7 | 3 | 0
Not completed — Failed to meet screening requirements. | 7 | 3 | 0
Period: Induction Treatment With Y90
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Started | 8 | 9 | 0
Completed | 8 | 9 | 0
Not Completed | 0 | 0 | 0
Period: Cycle 1 (DLT Monitoring Period)
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Started | 8 | 9 | 0
Received Nivolumab Dose | 6 | 7 | 0
Completed | 6 | 6 | 0
Not Completed | 2 | 3 | 0
Not completed — Progressive Disease | 2 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Cycle 2 and Beyond
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Started | 6 | 6 | 0
Completed | 5 | 6 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: 2 Year Follow-up
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Started | 6 (All patients who receive at least one dose of nivolumab go into follow-up.) | 7 (All patients who receive at least one dose of nivolumab go into follow-up.) | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 7 | 0
Not completed — Death | 6 | 7 | 0

BASELINE CHARACTERISTICS:
Population: Although the MTD was determined at dose level 2 (240 IV every 2 weeks), Phase 1b never opened for accrual due to funding issues. In Phase I dose lvl 1, 7 patients failed screening. In Phase I does lvl 2, 3 patients failed screening. Included here patients that were treated on study. 10 patients were screen fails (not treated) and not included here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks) | Total
Number analyzed (Participants) | 8 | 9 | 0 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 0 | 10
  >=65 years | 4 | 3 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 0 | 7
  Male | 6 | 4 | 0 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 7 | 8 | 0 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 8 | 6 | 0 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 |  | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: To identify maximum tolerated dose (MTD) of nivolumab for combination treatment of nivolumab following Y-90 in patients with advanced hepatocellular carcinoma. The MTD will be defined as the highest dose of nivolumab that causes dose limiting toxicities (DLTs) in <2 of 6 patients. The Phase I portion of the study follows a 3+3 dose escalation design. Nivolumab has two dose levels: Level 1: 80mg IV every 2 weeks, Level 2: 240mg IV every 2 weeks. Toxicity will be assessed using the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), version 4.03. A DLT is defined as an Adverse Event (AE) or abnormal laboratory value assessed as at least possibly related to the study medication, occurs ≤ 28 days (1 cycle) following the first dose of nivolumab and meets any of the criteria listed in the Protocol (Section 4.3.1).
Time Frame: The first cycle of treatment with nivolumab (28 days)
Measure: Number; unit: mg of nivolumab, IV
Groups:
- Phase I (Yttrium Y 90 Glass Microspheres, Nivolumab): Patients in Phase I receive yttrium Y 90 glass microspheres IA. Approximately 4 weeks after yttrium Y 90 glass microspheres treatment, patients receive nivolumab IV over 30-60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Phase I follows a 3+3 dose escalation design. There are two dose levels of nivolumab, Level 1: 80mg IV every 2 weeks, and Level 2: 240mg IV every 2 weeks.
  Laboratory Biomarker Analysis: Correlative studies
  Nivolumab: Given IV
  Yttrium Y 90 Glass Microspheres: Given IA
Arm/Group | Phase I (Yttrium Y 90 Glass Microspheres, Nivolumab)
Number analyzed (Participants) | 12
mg of nivolumab, IV | 240

2. Primary Outcome: Phase IB: Objective Response Rate (ORR)
Description: Evaluate tumor response by assessing the proportion of patients with Objective response rate (ORR) (according to RECIST v. 1.1 criteria) to the combination treatment of nivolumab with Y-90 by examining imaging scans. Per RECIST v. 1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: At baseline and every 8 weeks for the first 13 months and then every 12 weeks up to 2 years
Population: Due to funding issues, Phase 1b of the study never opened to accrual.
Arm/Group | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Who Experience Adverse Events
Description: Safety and tolerability of toxicities (according to the NCCN CTCAE v4.03) and tolerability of nivolumab and y-90 in patients with advanced hepatocellular carcinoma as graded using CTCAE 4.03 that are grade 3 - 5 for patients determined to be evaluable for other endpoints. In general the following severity definitions are true:
  Mild (grade 1): the event causes discomfort without disruption of normal daily activities.
  Moderate (grade 2): the event causes discomfort that affects normal daily activities.
  Severe (grade 3): the event makes the patient unable to perform normal daily activities or significantly affects his/her clinical status.
  Life-threatening (grade 4): the patient was at risk of death at the time of the event. Fatal (grade 5): the event caused death.
Time Frame: During treatment where (1 Cycle = 28 days) the range of cycles attempted was 1-14 and up to 100 days following the last administration of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks)
Number analyzed (Participants) | 5 | 5
Participants
  Lymphocyte count decreased | 2 | 1
  Abdominal pain | 1 | 0
  Blood bilirubin increased | 1 | 0
  Alkaline phosphatase increased | 1 | 0
  Keratitis | 1 | 0
  Thromboembolic event | 1 | 0
  Aspartate aminotransferase increased | 0 | 1
  Hyperglycemia | 0 | 2
  Creatinine increased | 0 | 1
  Investigations (other) | 1 | 0

4. Secondary Outcome: Progression Free Survival (PFS) at 24 Weeks (6 Months)
Description: Evaluate the percentage of patients alive and progression free at 24 weeks. PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression assessment will be performed by investigator each time the patients has a radiologic evaluation after 8 weeks of treatment. In general Progressive Disease (PD) will be assessed using RECIST v1.1 and defined as: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm). (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 24 weeks (6 months)
Measure: Number; unit: percentage of patients
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks)
Number analyzed (Participants) | 5 | 5
percentage of patients | 40 | 40

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR will be determined at 24 weeks from the start of nivolumab treatment by the sum of complete response (CR), partial response (PR) and stable disease (SD) according to measurement of target and non-target lesions as assessed by RECIST v1.1 where generally the following definitions are true:
  CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm.
  PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study.
Time Frame: At 24 weeks (6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks)
Number analyzed (Participants) | 5 | 5
Participants | 4 | 4

6. Other Pre Specified Outcome: PD-L1 Protein Expression
Description: Tumor tissue will be used to examine expression of PD-L1 protein on tumor cells.
Time Frame: At baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Expression Level of Biomarker of Inflammatory/Immune Signature
Description: Evaluate biomarker expression level using immunohistochemistry or flow cytometry.
Time Frame: Up to 2 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Circulating Free DNA (cfDNA) Mutation Analyses
Description: Change in clonal burden landscape will be analyzed to investigate its correlation with treatment response or development of resistance to treatment.
Time Frame: Every 8 weeks for the first 24 weeks then every 16 weeks up to 2 years
Reporting Status: Not Posted

9. Post Hoc Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from start of treatment to time of death and is summarized using Kaplan-Meier product limit curve and estimates.
Time Frame: Followed during treatment (1 Cycle = 28 days the range of cycles attempted was 1-14) and for up to 2 years during follow up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks)
Number analyzed (Participants) | 5 | 5
months | 14.65 [8.77 to 14.65] | 4.50 [2.30 to 9.36]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 3 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment, where 1 Cycle = 28 days the range of cycles attempted was 1-14.
Description: Patients who signed consent/did not initiate treatment are included as at risk for SAE but not at risk for other AEs due to 1 out of 10 screenfail patients experiencing an SAE. All cause mortality and other adverse events are assessed from first dose of study treatment. Only patients that received at least 1 dose of study drug are included in all cause mortality and other adverse events. SAEs are assessed from patient signing consent.
Arm/Group | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks)
All-Cause Mortality (participants affected / at risk) | 7/8 | 9/9 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/15 | 9/12 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) (N=15) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) (N=12) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks) (N=0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 — One patient also experienced right lower extremity cellulitis at the time of the event.
Thromboembolic event (Vascular disorders) | 2 | 0 | 0 — * One patient also experienced keratits and influenza at the time of the event. * One patient also experienced hypoxia at the time of the event.
Hepatic Failure (Hepatobiliary disorders) | 1 | 0 | 0 — One patient also experienced fever, lethargy, and upper gastrointestinal hemorrhage at the time of the event.
Hepatic Encephalopathy (Hepatobiliary disorders) | 2 | 0 | 0
Spontaneous Bacterial Peritonitis (Infections and infestations) | 1 | 1 | 0 — One patient also experienced cognitive disturbance at the time of the event. One patient also experienced UTI and encephalopathy at the time of the event.
Sepsis (Infections and infestations) | 1 | 1 | 0 — One patient also experienced diarrhea at the time of the event. One patient also experienced fatigue and altered mental state at the time of the event.
Abdominal Distention (Gastrointestinal disorders) | 1 | 0 | 0 — One patient also experienced abdominal pain at the time of the event.
Fever (General disorders) | 1 | 0 | 0
Intracranial Hemorrhage (Nervous system disorders) | 1 | 0 | 0 — One patient also experienced aspiration at the time of the event.
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — One patient also experienced hypercalcemia at the time of the event.
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 — One patient also experienced gait disturbance at the time of the event.
Death NOS (General disorders) | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 — This patient failed screening and did not receive Y90 or nivolumab.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Nivolumab Dose Lvl 1 (80mg IV Every 2 Weeks) (N=8) | Phase I, Nivolumab Dose Lvl 2 (240mg IV Every 2 Weeks) (N=9) | Phase 1b at Nivolumab MTD (240mg IV, Every 2 Weeks) (N=0)
Anemia (Blood and lymphatic system disorders) | 4 | 6 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0
Blurred vision (Eye disorders) | 0 | 2 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 0
Ascites (Gastrointestinal disorders) | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Edema limbs (General disorders) | 3 | 3 | 0
Fatigue (General disorders) | 5 | 5 | 0
Fever (General disorders) | 2 | 1 | 0
Gait disturbance (General disorders) | 1 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 1 | 0
Localized edema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 3 | 0
Pain (General disorders) | 1 | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 3 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 6 | 0
Alkaline phosphatase increased (Investigations) | 6 | 6 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 7 | 0
Blood bilirubin increased (Investigations) | 6 | 9 | 0
Creatinine increased (Investigations) | 1 | 2 | 0
INR increased (Investigations) | 2 | 4 | 0
Investigations - Other, specify (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 7 | 7 | 0
Platelet count decreased (Investigations) | 4 | 5 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 0 | 3 | 0
White blood cell decreased (Investigations) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 5 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 6 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 7 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 5 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 4 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 2 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 3 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 2 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Hypertension (Vascular disorders) | 4 | 4 | 0
Hypotension (Vascular disorders) | 1 | 2 | 0
Thromboembolic event (Vascular disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
The total accrual goal of 40 patients was not met. Due to funding issues, Phase 1b of the study never opened to accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/29/NCT02837029/Prot_SAP_001.pdf